CLINICAL TRIAL: NCT06013839
Title: A Phase 2, Single-Arm, Open-Label, Multi-Center Study to Evaluate the Safety and Efficacy of TXA127/Angiotensin [1-7] in Non-Ambulant Patients With Duchenne Muscular Dystrophy (DMD) Cardiomyopathy Who Are Receiving Systemic Glucocorticoids
Brief Title: TXA127 in Non-Ambulant Patients With DMD Cardiomyopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Constant Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXA127-DMD-002
Record Dates: First submitted 2023-08-16; First posted 2023-08-28 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-09

CONDITIONS: DMD-Associated Dilated Cardiomyopathy
MeSH Terms: conditions — Dmd-Associated Dilated Cardiomyopathy | interventions — angiotensin I (1-7)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TXA127 SC 0.5mg/kg/day (Experimental): TXA127 (talfirastide) 0.5mg/kg/day given via subcutaneous injection for 6 months
  Interventions: Drug: talfirastide

INTERVENTIONS:
Drug: talfirastide — TXA127 (talfirastide) is a pharmaceutically formulated angiotensin (1-7) heptapeptide, identical to the endogenously produced, non-hypertensive derivative of angiotensin II (Ang II).
  Other Names: TXA127; Angiotensin-(1-7)

SUMMARY:
This open-label, single-arm multi-center study studying the safety and efficacy of TXA127 on non-ambulant patients with DMD Cardiomyopathy will comprise of two phases:

1. 6-month open-label treatment phase: Male DMD patients with documented cardiomyopathy, will receive a daily subcutaneous injection of TXA127 0.5 mg/kg. Treatment will be provided for 6 months. Treatment safety will be assessed by collection and review of AEs, vital signs, ECGs, physical examinations, PFTs, and laboratory parameters on Day 1, Month 1, and Month 6. Ejection Fraction, upper extremity strength and biomarker levels will be assessed at these study visits as well. In addition, an abbreviated safety visit will be conducted at Month 3.
2. 12-month optional extension phase: Patients will continue the same study drug regime for an additional 12 months. The primary objective of this phase is to obtain long-term safety data. Efficacy data will also be collected. Safety, efficacy, and exploratory biomarkers will be assessed at Month 12 and Month 18, using the same methods as in the treatment phase. In addition, abbreviated safety visits will be conducted at Month 9 and Month 15.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects 16 years of age or older who provide informed consent and can follow up with protocol procedures. Parental or guardian consent is required for subjects at least 16 years of age but younger than 18 years of age.
2. Documented diagnosis of Duchenne muscular dystrophy by genetic mutation analysis.
3. Documented cardiomyopathy, as assessed by echocardiogram with:

   1. For a patient ≤ 20 years of age, EF > 35% and < 55% and fractional shortening of ≤ 28% at the time of screening.
   2. For a patient > 20 years of age, EF > 20% and fractional shortening ≤ 28% at the time of screening.
4. Reproducible (+/- 10%) difference between screening and baseline of percent predicted FVC , using the best out of 3 efforts at each visit:

   1. For a patient ≤ 20 years of age, FVC between 45% and 85%, inclusive. Patient should not utilize non-invasive ventilation such as CPAP or BiPAP.
   2. For a patient >20 years of age, all of the following should exist: FVC > 20%, EF > 20% in baseline ECHO and ability to be off non-invasive ventilation, such as CPAP and BiPAP, for at least 4 consecutive hours a day (24 hours period).
5. Subjects must be taking systemic glucocorticoids for at least six months prior to screening.
6. Subjects taking mineralocorticoid receptor antagonists, must be taking the drug for at least three months prior to screening
7. Non-ambulant and cared for by a trained caregiver

Exclusion Criteria:

1. Therapy with intravenous inotropic or vasoactive medications at the time of screening
2. Planned or likelihood of major surgery in the 6 months after planned enrollment.
3. Patient is using a left ventricular assist device (LVAD) or actively in the process of acquiring a LVAD.
4. Estimated glomerular filtration rate (GFR) <50 mL/min, as calculated by the CKD-EPI Creatinine equation 2021 (https://www.kidney.org/professionals/kdoqi/gfr_calculator)
5. Patient is suffering from unstable systemic allergic reaction(s), connective tissue disease or autoimmune disorder(s), requiring active intervention
6. History of cardiac tumor or current cardiac tumor
7. Known moderate-to-severe aortic stenosis/insufficiency or severe mitral stenosis/regurgitation
8. Current alcohol or drug abuse
9. Known history of chronic viral hepatitis unless considered cured based on hepatitis C RNA negative results
10. Hepatic dysfunction upon screening evidenced by bilirubin levels or gamma-GT levels above normal, deemed as clinically significant by the PI/Sub-I, and/or abnormal hematology (hematocrit <25%, WBC <3000/μl, platelets <100,000/μl), without a reversible, identifiable cause. Total bilirubin elevations > 2 times the upper reference range, consistent with Gilbert's Syndrome, may be enrolled if there is no other evidence of liver dysfunction
11. Uncontrolled diabetes (HbA1c >9.0 percent)
12. Inability to comply with protocol-related procedures, including required study visits
13. Any condition or other reason that, in the opinion of the investigator or Medical Monitor, would render the subject unsuitable for the study
14. Currently receiving or received within 90 days of enrollment (Day 1) an investigational treatment on another clinical study or expanded access protocol. This will include patients currently being treated or who have not completed follow-up to treatment with an investigational cell-based therapy within 6 months prior to enrollment and patients actively receiving an investigational therapy for cardiovascular repair/regeneration.

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of TXA127 in patients with DMD | 6 months plus 12 month extension
  Incidence of adverse events (AEs), their severity and relationship to treatment
To evaluate the effects of treatment on ejection fraction (EF) | 6 months plus 12 month extension
  Percent change in EF, as measured by echocardiogram (ECHO); Absolute change in EF, as measured by echocardiogram

SECONDARY OUTCOMES:
To evaluate the effects of treatment on upper extremity muscle function | 6 months plus 12 month extension
  Percent change in upper extremity strength, as measured by grip strength with a dynamometer; Absolute change in upper extremity strength, as measured by grip strength with a dynamometer
To evaluate the effects of treatment on fractional shortening (FS) | 6 months plus 12 month extension
  Percent and absolute change in fractional shortening as measured by echocardiogram

OTHER OUTCOMES:
To evaluate the effects of treatment on exploratory DMD-related clinical signs, FVC | 6 months plus 12 month extension
  Forced Vital Capacity (FVC) % predicted
  Absolute and percent (where applicable) change in the following biomarkers in the blood:
  * Troponin and Brain Natriuretic Peptide (BNP)
  * Brain-derived neurotrophic factor (BDNF)
To evaluate the effects of treatment on exploratory DMD-related clinical signs, PEF | 6 months plus 12 month extension
  Peak Expiratory Flow (PEF) % predicted (if available)
  Absolute and percent (where applicable) change in the following biomarkers in the blood:
  * Troponin and Brain Natriuretic Peptide (BNP)
  * Brain-derived neurotrophic factor (BDNF)
To evaluate the effects of treatment on exploratory DMD-related biomarkers, Troponin | 6 months plus 12 month extension
  Absolute and percent (where applicable) change in Troponin
To evaluate the effects of treatment on exploratory DMD-related biomarkers, BNP | 6 months plus 12 month extension
  Absolute and percent (where applicable) change in Brain Natriuretic Peptide (BNP)
To evaluate the effects of treatment on exploratory DMD-related biomarkers, BDNF | 6 months plus 12 month extension
  Absolute and percent (where applicable) change in Brain-derived neurotrophic factor (BDNF)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Franklin, MD, PhD, Study Chair — Constant Therapeutics LLC
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No